CLINICAL TRIAL: NCT01009333
Title: InterStim Therapy Programming Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1650
Record Dates: First submitted 2009-11-02; First posted 2009-11-06 (Estimated); Results first posted 2012-05-02 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Urgency Frequency; Urinary Urge Incontinence
Keywords: urgency frequency; urinary urge incontinence; InterStim Therapy
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low InterStim rate setting at 5.2 Hz (Experimental)
  Interventions: Device: InterStim Therapy at rate 5.2 Hz
- Medium InterStim rate setting at 14 Hz (Experimental)
  Interventions: Device: InterStim Therapy at rate 14 Hz
- High InterStim rate setting at 25 Hz (Experimental)
  Interventions: Device: InterStim Therapy

INTERVENTIONS:
Device: InterStim Therapy at rate 5.2 Hz — All subjects enrolled in this study were programmed to this rate setting for a 1-week period.
  Arms: Low InterStim rate setting at 5.2 Hz
Device: InterStim Therapy at rate 14 Hz — All subjects enrolled in this study were programmed to this rate setting for a 1-week period.
  Arms: Medium InterStim rate setting at 14 Hz
Device: InterStim Therapy — All subjects enrolled in this study were programmed to each rate setting (low, medium, high) for a 1-week period.
  Arms: High InterStim rate setting at 25 Hz

SUMMARY:
This study assessed the effect of different InterStim rate settings on voiding diary outcomes. Specifically, the study evaluated how 3 different rate settings affected the number of urinary incontinent episodes per day collected through a voiding diary. The study also evaluated how the 3 different rate settings affected other voiding diary measures including number of voids per day, degree of urgency before each void, number of pads used per day, and number of fecal incontinent episodes, questionnaires, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with either Neurostimulator Model 3023 (InterStim) or Neurostimulator Model 3058 (InterStim II) for at least 3 months - Implanted with tined lead models 3889 or 3093
* Tined lead is located in S2, S3, or S4
* Diagnosis before InterStim implant included urgency frequency (an average of 8 or more voids per day) and any amount of urinary urge incontinence over the voiding diary reporting period. The diary reporting period must be at least 2 days.
* Able to tolerate (ie, no complaint of pain or discomfort) acute high InterStim rate setting
* Able to tolerate (ie, no complaint of pain or discomfort) acute medium InterStim rate setting
* Able to tolerate (ie, no complaint of pain or discomfort) acute low InterStim rate setting
* Must be willing to maintain their current regimen (dosage and frequency) of any overactive bladder medication (anticholinergic or antimuscarinic) or tricyclic antidepression medication over the study duration
* Female subject 18 years of age or older
* Willing and able to accurately complete voiding diaries and questionnaires, attend visits, and comply with the study protocol that includes maintenance of InterStim programming settings over the course of the study.
* Able to consent to participate by signing the Informed Consent Form

Exclusion Criteria:

* Multiple sclerosis
* Reiter's syndrome
* Exclude diabetics unless the subject's diabetes is well-controlled with diet or medication
* History of spinal cord injury or a cerebral vascular accident (CVA)
* Active symptomatic urinary tract infection (UTI)
* Stress incontinence as the primary diagnosis
* Pelvic pain of uncertain etiology that is not associated with a voiding dysfunction or where pelvic pain is the primary complaint/diagnosis
* Interstitial cystitis as the primary diagnosis
* Urinary retention as the primary diagnosis
* Treatment of urinary symptoms with botulinum toxin in the past 12 months or any plan to have botulinum toxin treatment during the study
* Bilateral lead placement
* Have other implantable neurostimulator, pacemaker, or defibrillator
* Have knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or RF energy exposure
* Have an anticipated system modification within the next 1 month
* Women who are pregnant or planning to become pregnant or women of child-bearing potential who are not using a medically-acceptable method of birth control. Women of child-bearing age potential must undergo a pregnancy test, with a clear negative result, no more than 7 days prior to randomization visit.
* Subjects who frequently use the patient programmer to change device program settings. "Frequently" is defined as at least once a day and does not include shutting off the device for safety purposes.
* Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol
* Study site personnel will contact the Medtronic Study Manager to determine if a potential subject who plans to enroll in another investigational device or drug trial, or is currently enrolled in an investigational device or drug trial is eligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen McGuire, Ph.D., Study Director — MedtronicNeuro
Locations (1):
- Kenneth Peters, MD, Royal Oak, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Start at 5.2 Hz, Then 14 Hz, Then 25 Hz: Participants started with Low InterStim Rate Setting at 5.2 Hz, then progressed to Medium InterStim Rate Setting at 14 Hz, then High InterStim Rate Settings at 25 Hz until they completed all three settings.
- Start at 5.2 Hz, Then 25 Hz, Then 14 Hz: Participants started with Low InterStim Rate Setting at 5.2 Hz, then progressed to High InterStim Rate Setting at 25 Hz, then Medium InterStim Rate Settings at 14 Hz until they completed all three settings.
- Start at 14 Hz, Then 5.2 Hz, Then 25 Hz: Participants started with Medium InterStim Rate Setting at 14 Hz, then progressed to Low InterStim Rate setting at 5.2 Hz, then High InterStim Rate Settings at 25 Hz until they completed all three settings.
- Start at 14 Hz, Then 25 Hz, Then 5.2 Hz: Participants started with Medium InterStim Rate Setting at 14 Hz, then progressed to High InterStim Rate setting at 25 Hz, then Low InterStim Rate Settings at 5.2 Hz until they completed all three settings.
- Start at 25 Hz, Then 5.2 Hz, Then 14 Hz: Participants started with High InterStim Rate Setting at 25 Hz, then progressed to Low InterStim Rate setting at 5.2 Hz, then Medium InterStim Rate Settings at 14 Hz until they completed all three settings.
- Start at 25 Hz, Then 14 Hz, Then 5.2 Hz: Participants started with High InterStim Rate Setting at 25 Hz, then progressed to Medium InterStim Rate setting at 14 Hz, then Low InterStim Rate Settings at 5.2 Hz until they completed all three settings.
Period: Week 1
Arm/Group | Start at 5.2 Hz, Then 14 Hz, Then 25 Hz | Start at 5.2 Hz, Then 25 Hz, Then 14 Hz | Start at 14 Hz, Then 5.2 Hz, Then 25 Hz | Start at 14 Hz, Then 25 Hz, Then 5.2 Hz | Start at 25 Hz, Then 5.2 Hz, Then 14 Hz | Start at 25 Hz, Then 14 Hz, Then 5.2 Hz
Started | 2 | 3 | 2 | 2 | 2 | 2
Completed | 2 | 3 (1 participant did not progress to the second period due to a protocol violation.) | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 2
Arm/Group | Start at 5.2 Hz, Then 14 Hz, Then 25 Hz | Start at 5.2 Hz, Then 25 Hz, Then 14 Hz | Start at 14 Hz, Then 5.2 Hz, Then 25 Hz | Start at 14 Hz, Then 25 Hz, Then 5.2 Hz | Start at 25 Hz, Then 5.2 Hz, Then 14 Hz | Start at 25 Hz, Then 14 Hz, Then 5.2 Hz
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 3
Arm/Group | Start at 5.2 Hz, Then 14 Hz, Then 25 Hz | Start at 5.2 Hz, Then 25 Hz, Then 14 Hz | Start at 14 Hz, Then 5.2 Hz, Then 25 Hz | Start at 14 Hz, Then 25 Hz, Then 5.2 Hz | Start at 25 Hz, Then 5.2 Hz, Then 14 Hz | Start at 25 Hz, Then 14 Hz, Then 5.2 Hz
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Incontinent Episodes Per Day
Description: In a diary, subjects are asked to rate each urine leaking episode at 'None', 'Slight', 'Moderate' or 'Heavy'. The urinary incontinence was counted if there is any degree of leaking, from 'Slight' to 'Heavy'. The total number of urinary incontinence was calculated per day.
Time Frame: three weeks
Population: Data from 12 subjects who completed the study were included in the efficacy analysis; data from 1 subject was excluded because the subject was not compliant with the study protocol and was subsequently withdrawn from the study. Data from all 13 subjects were used for safety reporting.
Measure: Mean (Standard Deviation); unit: Episodes Per Day
Arm/Group | Low InterStim Rate Setting at 5.2 Hz | Medium InterStim Rate Setting at 14 Hz | High InterStim Rate Setting at 25 Hz
Number analyzed (Participants) | 12 | 12 | 12
Episodes Per Day | 3.83 (2.27) | 2.37 (1.83) | 2.82 (2.1)
Statistical Analysis 1: Comparison: Low InterStim Rate Setting at 5.2 Hz vs High InterStim Rate Setting at 25 Hz; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis

2. Secondary Outcome: Number of Voids Per Day
Description: In a diary, subjects are asked clarify each void as 'urine', 'fecal' or 'both'. Either 'urine' or 'both' are counted as void for this analysis. The total number of voids was calculated per day.
Time Frame: three weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Voids Per Day
Arm/Group | Low InterStim Rate Setting at 5.2 Hz | Medium InterStim Rate Setting at 14 Hz | High InterStim Rate Setting at 25 Hz
Number analyzed (Participants) | 12 | 12 | 12
Voids Per Day | 9.33 (2.08) | 9.36 (2.34) | 9.57 (2.28)
Statistical Analysis 1: Comparison: Low InterStim Rate Setting at 5.2 Hz vs High InterStim Rate Setting at 25 Hz; Test type: Superiority or Other; p = 0.589, Mixed Models Analysis

3. Secondary Outcome: Number of Pads Per Day
Description: In a diary, subjects are asked to provide number of pads they used per day.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: Pads Per Day
Arm/Group | Low InterStim Rate Setting at 5.2 Hz | Medium InterStim Rate Setting at 14 Hz | High InterStim Rate Setting at 25 Hz
Number analyzed (Participants) | 12 | 12 | 12
Pads Per Day | 2.61 (1.64) | 1.84 (1.43) | 1.94 (1.61)
Statistical Analysis 1: Comparison: Low InterStim Rate Setting at 5.2 Hz vs High InterStim Rate Setting at 25 Hz; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Low InterStim Rate Setting at 5.2 Hz | Medium InterStim Rate Setting at 14 Hz | High InterStim Rate Setting at 25 Hz
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/13 | 5/12 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low InterStim Rate Setting at 5.2 Hz (N=13) | Medium InterStim Rate Setting at 14 Hz (N=12) | High InterStim Rate Setting at 25 Hz (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Change in sensation of stimulation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Medtronic
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Painful defaecation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No